CLINICAL TRIAL: NCT00183235
Title: Effectiveness of Aripiprazole to Reduce Craving for Alcohol and Drinking Under Natural Observation, During Cue Induced Brain Imaging, and During a Motivated Free Choice Drinking Procedure Compared to Placebo
Brief Title: Aripiprazole Effects on Alcohol Reactivity and Consumption
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAANT010761-2005b; P50AA010761 (NIH); NIH P50 AA010761
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Alcoholism; Craving
MeSH Terms: conditions — Alcoholism | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole (up to 15 mg/day) for 8 days

SUMMARY:
The purpose of this study is to determine whether aripiprazole (marketed dopamine stabilizer) is effective in reducing of alcohol craving compared to placebo.

DETAILED DESCRIPTION:
Non-treatment seeking individuals meeting criteria for alcohol dependence (N=30) will be recruited through advertisement and paid for their participation. Alcoholics, after baseline evaluation, will be assigned through urn randomization to one of two experimental groups in which they will receive either aripiprazole (up to 15 mg/day) or an identical placebo. Subjects will take the study drug or placebo for 8 days (day 1-6 being the natural observation period). After a minimum of 24 hours of abstinence from alcohol (day 7-8) they will undergo an alcohol administration (priming dose) and motivated free choice drinking procedure (on day 8). Alcoholic subjects will receive a brief counseling session at the end of the study to enhance their awareness of problem drinking and to motivate them to seek treatment. Referral for treatment will be offered.

Each subject will undergo a functional MRI brain scan with cue stimulation on day 7, on the evening before the alcohol administration paradigm. fMRI brain imaging technology will be used to determine if alcoholics treated with aripiprazole differ in alcohol cue-induced activity in the nucleus accumbens. It is hypothesized that aripiprazole will reduce nucleus accumbens activation to alcohol cues compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 65
* Meets the DSM IV criterion for current alcohol dependence including "loss of control over drinking" (criterion 3 and/or 4).
* Currently is not engaged in, and does not want treatment for, alcohol related problems.
* Able to read and understand questionnaires and informed consent.
* Lives within 50 miles of the study site.
* Able to maintain abstinence for up to two days (without the aid of detox medications) as determined by self report and breathalyzer measurements.
* *Inclusion for fMRI imaging:

  * Does not have metal objects in the head/neck.
  * Does not have a history of claustrophobia leading to significant clinical anxiety symptoms.

Exclusion Criteria:

1. Currently meets DSM IV criteria for any other psychoactive substance dependence disorder.
2. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days as evidenced by self-report and urine drug screen. For marijuana - no use within the last seven days.
3. Meets DSM IV criteria for current axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders and eating disorders, any other psychotic disorder or organic mental disorder.
4. Has current suicidal ideation or homicidal ideation.
5. Need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications.
6. Current use of disulfiram.
7. Clinically significant medical problems such as, cardiovascular, renal, GI, or endocrine problem that would impair participation or limit medication ingestion.
8. Past history of alcohol related medical illness such as gastrointestinal bleeding, pancreatitis, peptic ulcer, hepatic cirrhosis or alcoholic hepatitis.
9. Hepatocellular disease indicated by elevations of SGPT (ALT) or SGOT (AST) greater than 2 1/2 times normal at screening.
10. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
11. Has current charges pending for a violent crime (not including DUI related offenses).
12. Does not have a stable living situation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
For the Efficacy Hypotheses, the primary dependent variables are
(First) "Natural" alcohol consumption period -- total number of drinks consumed during the 5-day observation period
(Second) Limited access alcohol consumption paradigm -- Total number of drinks consumed
(Third) Activation of nucleus accumbens after cue stimulation
For the Safety and Tolerability Hypotheses, the primary dependent variables are
(First) Number of drop-outs due to adverse events
(Second) Number of side effects on symptom checklist
(Third) Change in liver function as indicated by ALT, AST

SECONDARY OUTCOMES:
Blood alcohol levels after priming drink
Average BAES stimulation score
SHAS score after alcohol priming drink
Change in POMS sub-scale scores
Change in Epworth Sleepiness Scale
Differential effects on the Quality of Sleep Scale
Craving (OCDS) change between day 1 and 6
Craving after alcohol priming

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F. Anton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Center for Drug and Alcohol Programs, Medical University of South Carolina, Charleston, South Carolina, United States